CLINICAL TRIAL: NCT00047229
Title: A Phase II Study of G3139 in Combination With Doxorubicin in Advanced Hepatocellular Carcinoma
Brief Title: Oblimersen and Doxorubicin in Treating Patients With Advanced Hepatocellular Carcinoma (Liver Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-011; CDR0000257565 (Registry Identifier: PDQ (Physician Data Query)); NCI-5798
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — oblimersen; Doxorubicin

ARMS (1):
- G3139 in combination with Doxorubicin (Experimental)
  Interventions: Biological: oblimersen sodium; Drug: doxorubicin hydrochloride

INTERVENTIONS:
Biological: oblimersen sodium
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as doxorubicin use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of doxorubicin by making tumor cells more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of combining oblimersen with doxorubicin in treating patients who have locally advanced, recurrent, or metastatic hepatocellular carcinoma (liver cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oblimersen and doxorubicin in patients with advanced hepatocellular carcinoma or other incurable solid tumor (closed to accrual as of 11/7/03). (Phase I completed as of 1/16/04.)
* Determine the efficacy of this regimen, in terms of objective response rate, in these patients.
* Determine the toxicity of this regimen in these patients.
* Determine the time to progression, response duration, progression-free survival, median survival, and overall survival rates in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study. (Phase I completed as of 1/16/04.)

Patients receive oblimersen IV continuously on days 1-7 and doxorubicin IV over 5 minutes on day 5. Treatment repeats every 4 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oblimersen and doxorubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients*, including 6 patients with hepatocellular carcinoma (HCC), are treated at the recommended phase II dose. (Phase I completed as of 1/16/04.)

NOTE: *Other solid tumors closed to accrual as of 11/7/03; only accruing HCC patients

PROJECTED ACCRUAL: A total of 12-18 patients will be accrued for the phase I portion of this study within 6 months (phase I completed as of 1/16/04). A total of 30 patients will be accrued for the phase II portion of this study within 10-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically or cytologically confirmed hepatocellular carcinoma (HCC)

    * Locally advanced, recurrent, or metastatic
    * Not candidates for surgical/radical therapies
  * Other solid tumor that is incurable (closed to accrual as of 11/7/03)
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Target lesion may not be in a previously irradiated field unless subsequent progression was documented
* No ascites
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 2,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* AST no greater than 5 times upper limit of normal (ULN)
* Albumin greater than 3.5 g/dL
* No cirrhosis worse than Childs-Pugh class A

Renal

* Creatinine no greater than 1.25 times ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* LVEF normal by MUGA
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Good nutritional status
* No encephalopathy
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No prior allergic reactions to compounds of similar chemical or biological composition to oblimersen or doxorubicin
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 1 prior biologic therapy regimen for patients with HCC
* At least 4 weeks since prior biologic therapy

Chemotherapy

* Patients with HCC:

  * No prior systemic chemotherapy
  * Prior chemotherapy as part of localized chemoembolization therapy may be allowed (no more than 150 mg/m^2 for doxorubicin) if completed at least 8 weeks before study treatment
* All other patients (closed to accrual as of 11/7/03):

  * At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
  * No prior doxorubicin, epirubicin, or other anthracycline

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No more than 3,000 cGy to fields including substantial bone marrow

Surgery

* At least 8 weeks since prior surgery
* Prior liver transplant for HCC allowed

Other

* Recovered from all prior therapy
* At least 8 weeks since other locally ablative therapies
* No concurrent commercial or other investigational agents or therapies
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-10; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Rate of objective response (complete and partial) | Up to 280 days
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR. Objective response rate of >= 30% is considered active, and <10% is considered inactive.

SECONDARY OUTCOMES:
Stable disease rate | Up to 280 days
Duration of response | Up to 280 days
Progression-free survival rate | Up to 280 days
Median survival rate | Up to 280 days
Overall survival rate | Up to 280 days
Safety and tolerability | Up to 280 days

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (3):
- Canada (3):
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Knox JJ, Chen XE, Feld R, Nematollahi M, Cheiken R, Pond G, Zwiebel JA, Gill S, Moore M. A phase I-II study of oblimersen sodium (G3139, Genasense) in combination with doxorubicin in advanced hepatocellular carcinoma (NCI # 5798). Invest New Drugs. 2008 Apr;26(2):193-4. doi: 10.1007/s10637-007-9104-1. Epub 2007 Dec 4. No abstract available. PMID 18060598
- [Result] Knox JJ, Chen E, Feld R, et al.: A phase II trial of oblimersen sodium (G3139) in combination with doxorubicin (DOX) in advanced hepatocellular carcinoma (HCC). NCI protocol # 5798. [Abstract] J Clin Oncol 24 (Suppl 18): A-14072, 2006.
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00047229